CLINICAL TRIAL: NCT05994222
Title: Turkish Translation of State Mindfulness Scale for Physical Activity; Validity, Reliability, and Cultural Adaptation
Brief Title: State Mindfulness Scale for Physical Activity: Validity and Reliability
Status: Completed | Type: Observational
Sponsor: Istinye University (Other)
Responsible Party: Sponsor
Other Study IDs: 22-120
Record Dates: First submitted 2023-08-08; First posted 2023-08-16 (Actual); Last update posted 2023-09-06 (Actual); Status verified 2023-09

CONDITIONS: Physical Inactivity
Keywords: physical activity; mindfulness; cultural adaptation; validity; relability
MeSH Terms: conditions — Sedentary Behavior; Motor Activity

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Assessment Group — Evaluation forms will be applied to the participant who meets the inclusion criteria by face-to-face interview method. The sociodemographic information of the participants and the time taken to answer the questions in the questionnaires will vary according to each participants but will take approximately 45 minutes. The second interview will be conducted with the patients for test-retest application at 1-week intervals.

SUMMARY:
The American College of Sports Medicine (ACSM) states that physical activity is very important for healthy adults as it provides many health and psychological benefits. Physical activity is any bodily movement produced by skeletal muscles that increases energy expenditure. physical activity; It is an important health behavior that can have a positive impact on physical, cognitive, and social well-being. In the population of athletes who qualify as physically active, the focus is not on adapting to exercise or improving physical activity. However, the inability of athletes to maintain their lifelong physical activity levels after retirement can cause health problems. Because physical activity behavior patterns are lifelong, it is important to understand the factors that contribute to physical activity.

Conscious awareness; It is defined as a mindset in the form of being aware of the present moment with the features that do not judge, accept and avoid. Mindfulness is often said to require both purposeful attention and an accepting attitude. Intention is also considered an important part of awareness. There is increasing interest in the role of mindfulness in the emergence of positive health outcomes. One possible benefit of mindful practice is that it can lead to intrinsic motivation. Until recently, there was no good way to measure the specific experience of mindfulness during physical activity to support this recommendation. A new scale called the State Mindfulness Scale for Physical Activity has been developed to help researchers better understand how people feel about their physical activity.

The State Mindfulness Scale for Physical Activity is a 12-item scale to measure mindfulness during a specific physical activity. The scale is based on the Situational Conscious Awareness Scale, which measures objects (mental and physical) and the quality of situational conscious awareness. The original scale was not comprehensive enough to capture the full spectrum of physical experiences. The State Mindfulness Scale for Physical Activity was developed to assess different aspects of mindfulness (mental and physical) during physical activity to better understand the physical activity experience. There are six items that use awareness of objects of mental experience and six items that use awareness of objects of physical or physical experience. State Mindfulness Scale for Physical Activity has been successfully adapted to Spanish, Italian and Brazilian.

Despite the increase in Turkish assessment tools in the field of physical activity in recent years, psychological assessment tools are very few. The aim of this study is to translate, culturally adapt and validate the Turkish version of the State Mindfulness Scale for Physical Activity.

ELIGIBILITY:
Inclusion Criteria:

* Be a licensed athlete between the ages of 18 and 35
* Be literate in Turkish

Exclusion Criteria:

* Having an ongoing injury

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy volunteers aged 18-35
Sampling Method: Non-Probability Sample
Enrollment: 132 (Actual)
Dates: Start 2023-08-08 (Actual); Primary Completion 2023-08-30 (Actual); Study Completion 2023-09-02 (Actual)

PRIMARY OUTCOMES:
State Mindfulness Scale for Physical Activity | 2 weeks
  It was developed by Cox et al (2015). It is a 12-item scale used to measure conscious awareness during a specific physical activity. The scale is based on the State Mindfulness Scale for Physical Activity, which measures objects (mental and physical) and the quality of situational conscious awareness. The State Mindfulness Scale for Physical Activitywas developed to assess different aspects of mindfulness (mental and physical) during physical activity in order to better understand the physical activity experience. Six items use awareness of objects of mental experience and six items use awareness of objects of physical or physical experience.
Behavioral Regulations in Exercise Scale-2 | 2 weeks
  It consists of 19 items and five subscales. These are: external regulation, introjected regulation, defined regulation, internal regulation and amotivation subscales. The external regulation and internal regulation subscales consist of four items, while the introjected regulation and defined regulation subscales consist of three items. The unmotivated subscale consists of 4 items. It is a 5-point Likert-type scale with scores ranging from 0 to 4, consisting of "definitely not true", "sometimes true" and "definitely true".
International Physical Activity Questionnaire Short Form | 2 weeks
  In our study, the self-administered short form of the questionnaire with 7 questions covering the last 1 week will be used to evaluate the level of physical activity. Calculation of the total score of the short form includes the sum of time (minutes) and frequency (days) of walking, moderate-intensity activity, and vigorous activity. The sitting score is calculated separately. A score is obtained as "MET-minutes/week" by multiplying the minutes, days and MET values.

CONTACTS AND LOCATIONS:
Locations (1):
- Istinye University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No